CLINICAL TRIAL: NCT00118703
Title: A 4 Week Randomized, Double Blind, Placebo Controlled Study of GW685698X Aq Nasal Spray 100mcg QD in Adults and Adolescents With Vasomotor Rhinitis
Brief Title: Once-Daily Investigational Nasal Spray In Adults And Adolescents With Vasomotor Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR30007
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-03

CONDITIONS: Vasomotor Rhinitis; Rhinitis, Vasomotor
Keywords: nonallergic rhinitis; GW685698X; VMR; vasomotor rhinitis
MeSH Terms: conditions — Rhinitis, Vasomotor

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of GW685698X 100mcg once daily (QD) aqueous nasal spray with vehicle placebo nasal spray in adult and adolescent subjects (12 years of age and older) with vasomotor rhinitis (VMR).

ELIGIBILITY:
Inclusion criteria:

* Must be outpatients.
* Diagnosis of VMR (vasomotor rhinitis).
* Literate in English or native language.

Exclusion criteria:

* Significant concomitant medical condition.
* Use corticosteroids or other allergy medications during the study.
* Used tobacco products within the past year.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2005-07-01; Primary Completion 2006-02-01 (Actual); Study Completion 2006-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (38):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Blue Bell, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, South Burlington, Vermont
- Canada (4):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Germany (4):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Ponce, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR30007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The actual dose delivered from the product was 27.5 micrograms (µg) /actuation, which is therefore proposed as the label claim rather than 25 µg/actuation. Based on this spray content assessment, the dose examined in this study was actually 110 µg rather than the 100 µg dose indicated in the protocol.
Pre-assignment Details: Males and females >=12 years of age, diagnosed with vasomotor rhinitis (VMR) and meeting the symptom requirements entered a 7 to 14 days screening period. Following screening period, participants meeting specified symptom criteria received treatment of either fluticasone furoate or placebo in 1:1 ratio up to 4 weeks.
Groups:
- Placebo: Participants were instructed to self administer two sprays of placebo into each nostril once daily (QD) in the morning (ante meridian [AM]), following pre-dose symptom assessment. Administration of the dose was performed by alternately spraying one spray to each nostril followed by a second spray to each nostril.
- Fluticasone Furoate 110 µg QD: Participants were instructed to self administer two sprays of fluticasone furoate 110 µg into each nostril QD in the morning (AM), following pre-dose symptom assessment. Administration of the dose was performed by alternately spraying one spray to each nostril followed by a second spray to each nostril.
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD
Started | 173 | 174
Completed | 168 | 165
Not Completed | 5 | 9
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Participant took two different treatment | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were instructed to self administer two sprays of placebo into each nostril QD in the morning (AM), following pre-dose symptom assessment. Administration of the dose was performed by alternately spraying one spray to each nostril followed by a second spray to each nostril.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD | Total
Number analyzed (Participants) | 173 | 174 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (14.72) | 43.8 (15.44) | 43.9 (15.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 124 | 232
  Male | 65 | 50 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 164 | 167 | 331
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daily Reflective Total Nasal Symptom Scores (rTNSS)
Description: The TNSS was the sum of the individual symptom scores for rhinorrhoea, nasal congestion and post-nasal drip which was scored on a scale of 0-3 (total score 0-9). The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. The rTNSS was a rating of the severity of symptoms over the previous 12 hours and was performed in the morning (AM rTNSS) and evening (post meridian [PM] rTNSS). The daily rTNSS was the sum of two assessments. The Baseline daily rTNSS was defined as the average of the daily rTNSS over the 4 consecutive 24-hour periods prior to randomization, including the assessment on the morning of randomization. Change from Baseline was calculated as the on-treatment value minus the Baseline.
Time Frame: Baseline and up to Week 4
Population: Intent-to-Treat (ITT) population comprised of all participants who were randomized and received at least one dose of study drug. Only participants present at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD
Number analyzed (Participants) | 172 | 172
Score on a scale | -2.11 (0.15) | -2.01 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 µg QD; Test type: Superiority or Other; p = 0.604, ANCOVA; The analysis method was adjusted for Baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Final Values) = 0.094, 95% CI 2-sided [-0.26 to 0.45]

2. Secondary Outcome: Mean Change From Baseline in Morning (AM) Pre-dose Instantaneous Total Nasal Symptom Scores (iTNSS)
Description: The morning pre-dose iTNSS was the sum of the individual symptom score for rhinorrhoea, nasal congestion and postnasal drip performed immediately prior to taking the daily dose which were scored on a scale of 0-3 (total score 0-9). The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. The Baseline daily iTNSS was defined as the average of the daily iTNSS over the 4 consecutive 24-hour periods prior to randomization, including the assessment on the morning of randomization. Change from Baseline was calculated as the on-treatment value minus the Baseline value.
Time Frame: Baseline and up to Week 4
Population: ITT population. Only participants available at the specified timepoint were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD
Number analyzed (Participants) | 172 | 172
Score on a scale | -1.65 (0.14) | -1.59 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 µg QD; Test type: Superiority or Other; p = 0.729, ANCOVA; The analysis method was adjusted for Baseline iTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.29 to 0.41]

3. Secondary Outcome: Number of Participants Based on Overall Evaluation of Response to Therapy
Description: Participants were evaluated effectiveness of study medication for relieving non-allergic rhinitis symptoms over the entire treatment period. The overall evaluation of response to therapy was based on a 7-point categorical scale (1-7) where the participants rate their perception of the change or lack of change in their VMR symptoms at the end of the study. The 7 categories were: 1: significantly improved, 2: moderately improved, 3: mildly improved, 4: no change, 5: mildly worse, 6: moderately worse and 7: significantly worse. Effectiveness of study medication for relieving VMR symptoms over the entire treatment period.
Time Frame: Week 4 (Day 29) or Early Withdrawal
Population: ITT Population. Only participants available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD
Number analyzed (Participants) | 172 | 171
Participants
  Significantly Improved | 20 | 28
  Moderately Improved | 39 | 41
  Mildly Improved | 42 | 43
  No Change | 63 | 50
  Mildly Worse | 3 | 4
  Moderately Worse | 2 | 3
  Significantly Worse | 3 | 2
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 µg QD; Test type: Superiority or Other; p = 0.064, Regression, Logistic; Overall evaluation of response to therapy was illustrated and analyzed using logistic regression adjusting for age, gender, investigator, and treatmen

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from on or after the randomization date (Up to Day 34).
Description: ITT Population was used.
Arm/Group | Placebo | Fluticasone Furoate 110 µg QD
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/173 | 1/174
Other Adverse Events (participants affected / at risk) | 38/173 | 42/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=173) | Fluticasone Furoate 110 µg QD (N=174)
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=173) | Fluticasone Furoate 110 µg QD (N=174)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Headache (Nervous system disorders) | 16 | 14
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Nasopharyngitis (Infections and infestations) | 10 | 11
Upper respiratory tract infection (Infections and infestations) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.